CLINICAL TRIAL: NCT04200612
Title: The Therapeutic Effects of Equine-Assisted Psychotherapy on Lowering Aggression Levels Through an Increase of Emotion Regulation
Brief Title: The Therapeutic Effects of Equine-Assisted Psychotherapy
Acronym: EAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chua Yi Rong Shawn (Other)
Collaborators: Nanyang Technological University (Other); Therapeutic and Educational Riding in Singapore (THERIS) (Unknown)
Responsible Party: Sponsor-Investigator, Chua Yi Rong Shawn, Co-Investigator, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-19-357
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Aggression; Stress; Psychopathy; Empathy
Keywords: Equine-Assisted Psychotherapy; Emotion Regulation; Aggression; Outcomes; Randomized-Controlled Trials
MeSH Terms: conditions — Aggression; Antisocial Personality Disorder; Emotional Regulation | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: The design of the experiment will be a single-blind Randomized Controlled Trial. Participants are randomly assigned to either an intervention group, an active-control group or a placebo-control group. Participants in the intervention group will go through the 5-week EAP program consisting of the clinical processing following some activities found in EAP manuals. Participants in the active-control group will undergo a 5-week program that only involves interactions with horses without any clinical input (i.e. commonly coined as animal-assisted activities). Participants in the placebo-control group will undergo a 5-week movie screening of 1 hour each session that is related to horses in the lab.
Who Masked: Participant
Masking Description: Participants are informed that they will be randomly assigned to either a EAP horse interaction group or a EAP horse movie group. They are told that this study is meant to investigate the outcomes of two different types of EAP. In actuality, there are 3 groups in total - one intervention and two control groups. Participants in the intervention and active-control group will be told that they are in the EAP horse interaction group whereas participants in the placebo-control group are told that they are in the EAP horse movie group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): Participants in the intervention group will go through the 5-week EAP program consisting of the clinical processing following some activities found in EAP manuals.
  Interventions: Behavioral: Equine-Assisted Psychotherapy; Behavioral: Equine-Assisted Activities
- Active-control group (Active Comparator): Participants in the active-control group will undergo a 5-week program that only involves interactions with horses without any clinical input (i.e. commonly coined as animal-assisted activities).
  Interventions: Behavioral: Equine-Assisted Activities
- Placebo-control group (Placebo Comparator): Participants in the placebo-control group will undergo a 5-week movie screening of 1 hour each session that is related to horses.
  Interventions: Other: Placebo-control group

INTERVENTIONS:
Behavioral: Equine-Assisted Psychotherapy — Equine-Assisted Psychotherapy (EAP) involves working on the psychological goals set between the client and the mental health professional. This is done through the experiential interactions between the clients and the horse. This experiential aspect is vital as it allows clients to process the emotions, thoughts and behaviors that were expressed during sessions with the horse.
  Other Names: Equine-Facilitated Psychotherapy
  Arms: Intervention Group
Behavioral: Equine-Assisted Activities — Simple interactions with the horses that does not necessarily involve any goals being set between the client and the personnel handling the session. These can involve activities such as grooming or petting of the horse.
  Arms: Active-control group; Intervention Group
Other: Placebo-control group — This group will only be watching movies related to horses and they are told that this is another form of EAP even though this is not the case. This type of intervention has not been known to provide any therapeutic effect relevant to the study and thus is used as the placebo-control.
  Arms: Placebo-control group

SUMMARY:
Equine-assisted interventions (EAI) are an emerging form of alternate psychotherapy that has been increasingly found to produce improvements in various treatment outcomes. However, the paucity of randomized-controlled trials (RCTs) in the EAI literature prevents any definitive conclusions to be made about the general effectiveness of EAI. This study tests whether one form of EAI, Equine-Assisted Psychotherapy (EAP), reduces aggression and alters risk factors associated with aggression in young adults, and whether emotion regulation mediates any effect of EAP on aggression. In a single-blind RCT, undergraduate students will be randomly assigned to either an intervention group, an active-control group, or a placebo-control group. Participants in the intervention group will undergo a 5-week EAP program consisting of structured, interactive activities with horses followed by a clinical processing component. Participants in the active control group will undergo a 5-week program that only involves interactions with horses without any clinical input (i.e. commonly coined as animal-assisted activities). Participants in the placebo-control group will undergo 5 weeks of 1-hour movie sessions related to horses. There will be three waves of data collection measuring key outcome variables - t1 before the 1st session, t2 after the 3rd session, and t3 after the final session. Participants will complete questionnaires assessing the key outcomes of aggression, emotional well-being and academic performance. Other risk factors of antisocial behaviour such as psychopathy, level of empathy, emotion regulation and executive functioning will also be measured. To the author's knowledge, the current study is the first in Singapore to investigate if EAP can lower aggression levels and alter psychological risk factors for aggression in healthy young adults. In turn, these results could help inform the utility and validity of EAP in the forensic populations.

DETAILED DESCRIPTION:
The EAP program will span over the duration of 5 weeks, each week having a 1-hour session. 50 minutes will be allocated to interacting with the horses and the activities while the remaining 10 minutes will be allocated to the clinical processing of the behavior, thoughts and emotions that are observed during the session. This processing will be guided by trained therapists who hold the relevant qualifications (i.e. equine-assisted psychotherapy certification). 2 horses (an Oldenburg and a pony, aged 19 and 14 respectively), 2 therapists, and 2 experienced horse handlers will be present throughout the sessions. Each 1-hour session will consist a maximum of 8 participants that will be split into two groups of 4 such that 1 horse, 1 therapist and 1 experienced horse handler are attached to them.

The design of the experiment will be a single-blind Randomized Controlled Trial. Participants will be told that this study aims to investigate the therapeutic effects of two different EAP programs (either watching video clips related to horses or actual interactions with horses) and that they will be randomly assigned to either one. In actuality, participants are randomly assigned to either an intervention group, an active-control group or a placebo-control group. 3 time points of data collection are measured throughout the 5-week duration - t1 before the 1st session, t2 after the 3rd session, and t3 after the final session. All participants will go through the same questionnaire administered at each time point during the 5-week duration regardless of their assigned group. Participants in the intervention group will go through the 5-week EAP program consisting of the clinical processing following some activities found in EAP manuals. Participants in the active-control group will undergo a 5-week program that only involves interactions with horses without any clinical input (i.e. commonly coined as animal-assisted activities). Participants in the placebo-control group will undergo a 5-week movie screening of 1 hour each session that is related to horses in the lab.

Participant recruitment will begin as soon as possible once approval has been given and should not take longer than 2 weeks to recruit a total of 120 undergraduate students from both NUS and NTU.

The 5-week intervention program will be briefly structured as such:

Session 1: Introduction to grooming and horse safety This introductory session is aimed at getting participants to be familiar with the safety features when working with these horses as well as to be attentive to the warning cues that horses display that is indicative of their mood. Once that has been briefed, participants will be taught how to groom the horse as part of learning natural horsemanship skills. These includes brushing and cleaning the hooves of the horse.

Session 2: Review of grooming, learning to put on halter and leading the horse The second session is built upon the previous session in that reviews of grooming and horse safety will continually be surfaced throughout the program as such lessons is always an ongoing process. On top of that, participants will be taught how to put on a halter on the horse and to lead the horse. The session ends with a modified activity called Catch and Release which allows participants to have personal interaction with the horse.

Session 3: Review of grooming and Give-and-Take The third session is more focused on the importance of proper communication as this helps convey the investigators intentions across with greater accuracy while still remaining respectful and mindful of the other party on the receiving end. After the grooming segment, participants will engage in an activity called Give-and-Take which work improving communication in a non-verbal manner only through the string they are provided with to guide the horse.

Session 4: Review on grooming and Life's Little Obstacles This session is aimed at utilizing participants' critical thinking skills to achieve the objective of the activity. This is meant to push participants' out of their comfort zones which could bring about feelings of frustration and worry that can be processed after the activity is over. The activity that is meant to create such a roadblock is the Life's Little Obstacles whereby participants are told to make the horse jump over a low obstacle with multiple restrictions.

Session 5: Review on grooming, Equine Billiards, and closing This final session is aimed at utilizing participants' problem-solving skills through the use of non-verbal communication. This is done using the Equine Billiards activity whereby the lessons learnt from previous sessions would culminate in this one task. Following the processing of the activity after it ends, the therapy team and participants would gather in a circle for the program closure to integrate whatever they have learnt from the past 5-weeks.

GPower 3.1 was used to calculate an appropriate sample size for a medium effect size of 0.15, power at 0.95 and alpha error probability at 0.05. For a multiple linear regression analysis with 2 tested predictors and total number of 4 predictors, the calculation yielded a total sample size of 119. This number was rounded up to 120.

All data will be analyzed using SPSS version 22. Some potential analyses include multiple linear regression, ANCOVAs and their respective post-hoc t-tests, paired-sample t-tests to demonstrate significant changes between pre and post intervention groups, and PROCESS Macro for the mediator analysis.

ELIGIBILITY:
Inclusion Criteria:

* Do not have any medical allergies or discomfort from interaction with horses.

Exclusion Criteria:

* Participants who self-report an existing diagnosis for a psychological disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition: DSM-V

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Young Adult Behavioral Scale (YABS) | Immediately before the 1st intervention session
  Min. Value: 1 (never), Max. Value: 5 (always), higher scores indicate a higher likelihood in the domains of relational aggression, social aggression and interpersonal maturity.
Young Adult Behavioral Scale (YABS) | Immediately after the 3rd intervention session
  Min. Value: 1 (never), Max. Value: 5 (always), higher scores indicate a higher likelihood in the domains of relational aggression, social aggression and interpersonal maturity.
Young Adult Behavioral Scale (YABS) | Immediately after the 5th intervention session
  Min. Value: 1 (never), Max. Value: 5 (always), higher scores indicate a higher likelihood in the domains of relational aggression, social aggression and interpersonal maturity.
Reactive-Proactive Aggression Questionnaire (RPQ) | Immediately before the 1st intervention session
  Min. Value: 0 (never), Max. Value: 2 (often), higher scores indicate higher general aggression levels
Reactive-Proactive Aggression Questionnaire (RPQ) | Immediately after the 3rd intervention session
  Min. Value: 0 (never), Max. Value: 2 (often), higher scores indicate higher general aggression levels
Reactive-Proactive Aggression Questionnaire (RPQ) | Immediately after the 5th intervention session
  Min. Value: 0 (never), Max. Value: 2 (often), higher scores indicate higher general aggression levels
Depression Anxiety Stress Scale - 21 items (DASS-21) | Immediately before the 1st intervention session
  Min. Value: 0 (did not apply to me at all), Max. Value: 3 (applied to me very much, or most of the time), higher scores indicate poorer emotional well-being
Depression Anxiety Stress Scale - 21 items (DASS-21) | Immediately after the 3rd intervention session
  Min. Value: 0 (did not apply to me at all), Max. Value: 3 (applied to me very much, or most of the time), higher scores indicate poorer emotional well-being
Depression Anxiety Stress Scale - 21 items (DASS-21) | Immediately after the 5th intervention session
  Min. Value: 0 (did not apply to me at all), Max. Value: 3 (applied to me very much, or most of the time), higher scores indicate poorer emotional well-being
Motivated strategies for Learning Questionnaire (MSLQ) | Immediately before the 1st intervention session
  Min. Value: 1 (not at all true of me), Max. Value: 7 (very true of me), higher scores indicate greater motivations to learn using the different strategies
Motivated strategies for Learning Questionnaire (MSLQ) | Immediately after the 3rd intervention session
  Min. Value: 1 (not at all true of me), Max. Value: 7 (very true of me), higher scores indicate greater motivations to learn using the different strategies
Motivated strategies for Learning Questionnaire (MSLQ) | Immediately after the 5th intervention session
  Min. Value: 1 (not at all true of me), Max. Value: 7 (very true of me), higher scores indicate greater motivations to learn using the different strategies
Emotion Regulation Questionnaire (ERQ) | Immediately before the 1st intervention session
  Min. Value: 1 (strongly disagree), Max. Value: 7 (strongly agree), higher scores indicate greater likelihood of using the two types of emotion regulation strategies
Emotion Regulation Questionnaire (ERQ) | Immediately after the 3rd intervention session
  Min. Value: 1 (strongly disagree), Max. Value: 7 (strongly agree), higher scores indicate greater likelihood of using the two types of emotion regulation strategies
Emotion Regulation Questionnaire (ERQ) | Immediately after the 5th intervention session
  Min. Value: 1 (strongly disagree), Max. Value: 7 (strongly agree), higher scores indicate greater likelihood of using the two types of emotion regulation strategies
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | Immediately before the 1st intervention session
  Min. Value: 1 (almost never), Max. Value: 5 (almost always), higher scores indicate greater difficulties with emotion regulation
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | Immediately after the 3rd intervention session
  Min. Value: 1 (almost never), Max. Value: 5 (almost always), higher scores indicate greater difficulties with emotion regulation
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | Immediately after the 5th intervention session
  Min. Value: 1 (almost never), Max. Value: 5 (almost always), higher scores indicate greater difficulties with emotion regulation

SECONDARY OUTCOMES:
Self-Report Psychotherapy - Short Form (SRP-SF) | Immediately before the 1st intervention session
  Min. Value: 1 (strongly disagree), Max. Value: 5 (strongly agree), higher scores indicate higher levels of psychopathy
Self-Report Psychotherapy - Short Form (SRP-SF) | Immediately after the 3rd intervention session
  Min. Value: 1 (strongly disagree), Max. Value: 5 (strongly agree), higher scores indicate higher levels of psychopathy
Self-Report Psychotherapy - Short Form (SRP-SF) | Immediately after the 5th intervention session
  Min. Value: 1 (strongly disagree), Max. Value: 5 (strongly agree), higher scores indicate higher levels of psychopathy
Cognitive, Affective and Somatic Empathy Scales (CASES) | Immediately before the 1st intervention session
  Min. Value: 0 (rarely), Max. Value: 2 (often), higher scores indicate higher levels of empathy
Cognitive, Affective and Somatic Empathy Scales (CASES) | Immediately after the 3rd intervention session
  Min. Value: 0 (rarely), Max. Value: 2 (often), higher scores indicate higher levels of empathy
Cognitive, Affective and Somatic Empathy Scales (CASES) | Immediately after the 5th intervention session
  Min. Value: 0 (rarely), Max. Value: 2 (often), higher scores indicate higher levels of empathy
Trail Making Task - Part B (TMT - Part B) | Immediately before the 1st intervention session
  Unit of measure: Reaction Time (s), higher scores indicate higher levels of executive functioning, more specific to attention span and attentional task switching abilities
Trail Making Task - Part B (TMT - Part B) | Immediately after the 3rd intervention session
  Unit of measure: Reaction Time (s), higher scores indicate higher levels of executive functioning, more specific to attention span and attentional task switching abilities
Trail Making Task - Part B (TMT - Part B) | Immediately after the 5th intervention session
  Unit of measure: Reaction Time (s), higher scores indicate higher levels of executive functioning, more specific to attention span and attentional task switching abilities

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Choy, PhD, Principal Investigator — Nanyang Technological University; Lim SM Matthew, PhD, PsyD, Principal Investigator — National University of Singapore
Locations (1):
- Therapeutic and Educational Riding in Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
There is no plans for such sharing as of now.